CLINICAL TRIAL: NCT03954392
Title: Social Cognitive Training to Enhance the Efficacy of CBT for Depression in Youth: A Developmental Approach
Brief Title: CBT Enhanced With Social Cognitive Training
Acronym: CBT+SCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Judith Garber, Professor, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R61MH115125 (NIH); 1R61MH115125-01A1 (NIH)
Record Dates: First submitted 2019-05-15; First posted 2019-05-17 (Actual); Results first posted 2023-03-28 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-02

CONDITIONS: Depression
Keywords: Depression; Adolescents; Treatment
MeSH Terms: conditions — Depression | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: The study has two intervention arms: (1) CBT + SCT is cognitive behavioral therapy enhanced with training in social cognitive abilities (e.g., social perspective taking), and (2) CBT-only is cognitive behavioral therapy without the additional SCT training component. Adolescents are randomized to either condition. We will stratify randomization by gender, age (12-14; 15-17), race/ethnicity (minority status), and medication use.
Who Masked: Outcomes Assessor
Masking Description: The individuals who conduct the assessments of the outcome measures will be unaware of to which condition the participant was randomized
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBT+SCT (Experimental): Cognitive behavioral therapy plus social cognitive skills training (SCT)
  Interventions: Behavioral: Cognitive behavior therapy with social cognitive training (CBT+SCT)
- CBT-only (Active Comparator): Cognitive behavioral therapy only (without SCT)
  Interventions: Behavioral: CBT-only

INTERVENTIONS:
Behavioral: Cognitive behavior therapy with social cognitive training (CBT+SCT) — The cognitive behavioral therapy is based on Beck's cognitive therapy model for the treatment of depression. We will conduct individual therapy based on the Coping with Stress manual used in other depression treatment studies with adolescents. In addition, the investigators will teach the teen explicitly about theory of mind and social perspective taking during each session and we will use examples from their own life to help them learn the skills.
  Arms: CBT+SCT
Behavioral: CBT-only — The cognitive behavioral therapy is based on Beck's cognitive therapy model for the treatment of depression. The investigators will conduct individual therapy based on the Coping with Stress manual used in other depression treatment studies with adolescents.
  Arms: CBT-only

SUMMARY:
Depression in youth is a serious public health concern for which more personalized treatments are needed. This study will test the effect of an intervention aimed at enhancing depressed children's social cognitive capacities (e.g., ability to take another's perspective), thereby making treatment of depression in youth more efficient and effective. Participants in both the R61 (N=42) and R33 (N=82) will be youth between 12 and 17 years old currently experiencing a depressive disorder. Youth will be randomized to either an enhanced CBT intervention that teaches social cognitive skills, particularly social perspective taking and theory of mind as compared to CBT only. The primary target is improvement in the social cognitive skills at post treatment in the first trial (R61) and improvements in both social cognitive skills and depressive symptoms at post-treatment and at a 4-month follow-up (R33).

DETAILED DESCRIPTION:
Depression in youth is a recurrent and impairing disorder. Although some treatments have shown modest effects in children and adolescents (e.g., cognitive behavioral therapy -- CBT), there remains a critical need to build upon these therapies in order to reach even more youths with depression. One variable hypothesized to affect children's interpersonal relationships is their level of social cognitive development on abilities particularly relevant to social functioning and CBT (e.g., social perspective taking; theory of mind). The first RCT (R61) will test the efficacy of an intervention aimed at increasing children's social cognitive (SC) abilities.Youth (ages 12-17; N=42) with depression diagnoses or clinical levels of depressive symptoms (CESD > 20) will be randomized to either the social cognitive training enhanced CBT (SCT-CBT) or CBT only. Pre- and post-treatment evaluations will assess the social cognitions. In the second RCT (R33), we will conduct a replication trial with a new sample of 82 youth (ages 12-17) again randomized to SCT-CBT or CBT only. Youth will be evaluated with regard to the SC abilities (i.e., theory of mind), level of depressive symptoms, and social functioning at baseline, post-treatment, and at a 4-month follow-up (R33). Finally, in the R33 we will test if increases in SC abilities partially account for the relation between treatment condition and decreases in depression. If the SCT-CBT intervention significantly improves children's SC abilities and social functioning and decreases depression, then this will provide therapists with a more efficient and personalized treatment of depression in youth,

ELIGIBILITY:
Inclusion Criteria:

* 12- to 17-years-old
* diagnosis of a current depressive disorder (e.g., major depressive episode; persistent depressive disorder) or a score on the Children's Depression Rating Scale (CDRS) >= 40

Exclusion Criteria:

* ever met criteria for a diagnosis of bipolar disorder, schizophrenia, autism, or conduct disorder
* current alcohol or substance use disorder with significant impairment
* imminent risk of suicide
* reading level < 4th grade
* estimated IQ<80

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2019-02-11 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judy Garber, PhD, Principal Investigator — Vanderbilt University
Locations (2):
- United States (2):
  - Judy Garber, Nashville, Tennessee
  - Vanderbilt University, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was primarily through a university listserv
Pre-assignment Details: Participants were randomized to condition shortly after eligibility was confirmed.
Period: Overall Study
Arm/Group | CBT+SCT | CBT-only
Started | 23 | 22
Completed | 23 | 22
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CBT+SCT | CBT-only | Total
Number analyzed (Participants) | 23 | 22 | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 23 | 22 | 45
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.87 (1.49) | 14.82 (1.62) | 14.845 (1.545)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 14 | 29
  Male | 8 | 8 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 21 | 20 | 41
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 3 | 5
  White | 19 | 18 | 37
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 23 | 22 | 45
Faux Pas Recognition Test [Mean (Standard Deviation); unit: units on a scale] — The Faux Pas Recognition Task consists of 10 Faux Pas Stories and 10 Control Stories without a faux pas, scoring one point for every correct faux pas perception. The higher score is 20 and lower score 0, domain scores are scaled in a positive direction (i.e. higher scores denote higher theory of mind). The Faux Pas recognition task is individually administered by trained staff.
  units on a scale | 0.853 (0.083) | 0.851 (0.072) | 0.852 (0.077)
Children's Depression Rating Scale [Mean (Standard Deviation); unit: units on a scale] — The Children's Depression Rating Scale-Revised (CDRS-R) total score ranges from 17 (minimal or no depression symptoms) to 133 (indicates depression) is a semi-structured, clinician-rated instrument for use with youth between the ages of 6 to 17 years of age and their caregivers. The CDRS-R evaluates the presence and severity of symptoms commonly associated with depression in childhood. The scale measures 17 depressive symptoms, of which 3 are rated 1-5 and 14 are rated 1-7 (1 = no symptom difficulties; 5 or 7 = severe clinically significant difficulties) for a total score range of 17-113.
  units on a scale | 48.26 (5.66) | 48.77 (6.32) | 48.52 (5.98)

OUTCOME MEASURES:

1. Primary Outcome: Faux Pas Recognition Test
Description: The Faux Pas Recognition Task consists of 10 Faux Pas Stories and 10 Control Stories without a faux pas, scoring one point for every correct faux pas perception. The higher score is 20 and lower score 0; domain scores are scaled in a positive direction (i.e. higher scores denote higher theory of mind). Faux Pas Recognition test measures the ability to identify and explain faux pas situations where a character unintentionally insults another person due to lack of knowledge about some key feature of the other character.
Time Frame: week 12
Population: Participants were 45 youth (64% female), ages 12 through 17 years old (Mean = 14.84, S.D. = 1.54). Youth either met diagnostic criteria for a major depressive episode or persistent depressive disorder or a score of 35 or greater on the Children's Depression Rating Scale.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CBT+SCT | CBT-only
Number analyzed (Participants) | 23 | 22
score on a scale | 0.901 (0.059) | 0.854 (0.071)
Statistical Analysis 1: Comparison: CBT+SCT vs CBT-only; Statistical analysis will compare the post-intervention scores on the primary outcome (Faux Pas Recognition Test scores), controlling for pre-intervention scores; Test type: Other; p < 0.05, ANCOVA; Only one statistical test was conducted, therefore no adjustments for multiple comparisons was needed

2. Secondary Outcome: Children Depression Rating Scale - Revised
Description: The Children's Depression Rating Scale-Revised (CDRS-R) total score ranges from 17 (minimal or no symptoms of depression) to 133 (indicative of depression). The CDRS-R is a semi-structured, clinician-rated instrument designed for use with children and adolescents between the ages of 6 to 17 years of age and their caregivers. The CDRS-R evaluates the presence and severity of symptoms commonly associated with depression in childhood. The scale measures 17 depressive symptoms, of which 3 are rated 1-5 and 14 are rated 1-7 (1 = no symptom difficulties; 5 or 7 = severe clinically significant difficulties) for a total score range of 17-113. Scores above 35 are considered to represent clinically significant symptoms. We measured depressive symptoms with the CDRS-R as a secondary outcome.
Time Frame: week 12
Population: Study participants
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CBT+SCT | CBT-only
Number analyzed (Participants) | 23 | 22
score on a scale | 23.74 (5.59) | 34.59 (10.60)
Statistical Analysis 1: Comparison: CBT+SCT vs CBT-only; Test type: Other; p < 0.05, ANCOVA

ADVERSE EVENTS:
Time Frame: The period of time over which adverse event data were collected was baseline to 2.5 years. For each participant, the time frame was baseline through their study completion (about 14 weeks).
Description: The definition used to collect adverse event information was from the clinicaltrials.gov Definitions.
Arm/Group | CBT+SCT | CBT-only
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/22
Other Adverse Events (participants affected / at risk) | 0/23 | 0/22

LIMITATIONS AND CAVEATS:
COVID19 started during the trial. We were able to move to conducting the study remotely (e.g., Zoom). That is, assessments and therapy sessions were conducted on Zoom. Overall, moving to remote methods was not a problem and allowed us to continue the trial without disruption.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2019-06-02): https://cdn.clinicaltrials.gov/large-docs/92/NCT03954392/Prot_001.pdf
  • Statistical Analysis Plan (2019-06-02): https://cdn.clinicaltrials.gov/large-docs/92/NCT03954392/SAP_002.pdf
  • Informed Consent Form (2019-06-02): https://cdn.clinicaltrials.gov/large-docs/92/NCT03954392/ICF_003.pdf